CLINICAL TRIAL: NCT01823731
Title: A Pilot Test for Newly Developed Synoptic Operative Template for Ovarian Cancer (SOTOC): National Cancer Center - Peritoneal Carcinomatosis Index
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Yoon Park, Chief, Center for Uterine Cancer, National Cancer Center, Korea
Other Study IDs: NCCNCS-13-700
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: PCI,SOTOC, Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
objectives: To development of NCC-PCI-Operative Template (NPOT) for the objective description of perioperative tumor burden and surgical approaches in the management of ovarian cancer, tubal cancer, and primary peritoneal cancer

DETAILED DESCRIPTION:
* Informed consent
* Digital photography & Checking PCI (tumor size& location )
* Postoperative surveillance(tumor marker, image and physical examination)
* Developing the best fitting NCC-PCI template to reflect recurrence and survival pattern

ELIGIBILITY:
Inclusion Criteria:

* Preoperative clinical diagnosis of ovarian cancer, tubal cancer, and primary peritoneal carcinoma
* Available preoperative image study (CT and/or MRI and/or PET)
* Patients who gave a written informed consent
* Patients must be surgical candidate considering medical and psychological condition

Exclusion Criteria:

* Patients who refuse to participate or want to withdraw at anytime.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * ovarian cancer, tubal cancer, primary peritoneal cancer, mesothelioma, pseudomyxoma peritonei
  * Debulking operation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of Clinical Applicability about Synoptic Operative Template for Ovarian Cancer (SOTOC) | one year